CLINICAL TRIAL: NCT05436158
Title: The Use of a New Safe Angle Position for Implant Placement in the Anterior Region: A Cross-sectional Study
Brief Title: The Use of a New Safe Angle Position for Implant Placement in the Anterior Region.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Mohamed Fouad Shemais, Lecturer in the department of Oral Medicine & Periodontology, Cairo University
Other Study IDs: IDCE.N2
Record Dates: First submitted 2022-06-19; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Immediate Implant Placement; Esthetic Zone; Anterior Maxilla; Safe Angle Position
Keywords: Immediate dental implants; anterior maxilla; safe angle position

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Implant placement in the safe angle position in the anterior maxilla — After assessing the CBCT of patients, the immediate implants will be assessed if they were placed in the safe zone. the safe zone is described as; that there is an angle between the intersection of the incisal long axis perpendicular to the palate or the occlusal plane, and the long axis of the root. When this relation is shifted more palatal, where the incisal plane line will be at the cingulum position or slightly palatal to it, it is named the safe angle position. The more palatal relocation to the cingulum is performed according to the availability of palatal bone, the occlusion with the opposing dentition, the type of the restoration (screw vs cemented).

SUMMARY:
There is an angle between the intersection of the incisal long axis perpendicular to the palate or the occlusal plane, and the long axis of the root. When this relation is shifted more palatal, where the incisal plane line will be at the cingulum position or slightly palatal to it, it is named the safe angle position. The more palatal relocation to the cingulum is performed according to the availability of palatal bone, the occlusion with the opposing dentition, the type of the restoration (screw vs cemented).

The possibility of having a specific safe angle to place implants opens new interesting perspectives for immediate placement of dental implants.

The aim of the present study was to demonstrate how immediate implants in the safe angle position can be predictably achieve proper implant positioning, better esthetics and emergence profile as well as less stresses on the implant.

DETAILED DESCRIPTION:
Immediate implants are implants inserted immediately after surgical extraction of the teeth to be replaced. Creation of an anatomically correct emergence profile is one of the most important aspects in providing an esthetically pleasing implant-supported restoration. Dentists understand the risks involved when restored prostheses are subjected to non-axial loading. It has always been recommended to direct occlusal loads as close to the long axis of the fixture as possible. However, it is known that the loading on angled abutments is mostly off-axis, which raises the concern of how angled abutments generally perform with such an unfavourable loading regimen.

There is an angle between the intersection of the incisal long axis perpendicular to the palate or the occlusal plane, and the long axis of the root. When this relation is shifted more palatal, where the incisal plane line will be at the cingulum position or slightly palatal to it, it is named the safe angle position. The more palatal relocation to the cingulum is performed according to the availability of palatal bone, the occlusion with the opposing dentition, the type of the restoration (screw vs cemented).

The possibility of having a specific safe angle to place implants opens new interesting perspectives for immediate placement of dental implants.

The aim of the present study was to demonstrate how immediate implants in the safe angle position can be predictably achieve proper implant positioning, better esthetics and emergence profile as well as less stresses on the implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with immediate implants in the anterior region
2. Patient with preoperative and postoperative CBCT
3. Provide informed consent.

Exclusion Criteria:

1. patients without a preoperative CBCT.
2. 2- patients without an informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with immediate implants in the anterior region
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
presence of the implant in the safe angle | 6 months
  binary (Y/N) from CBCT
use of angled or straight abutment | 6 months
  Binary (straight/angled)

SECONDARY OUTCOMES:
Pink Esthetic Score | 6 months
  Pink Esthetic Score (1-14)

CONTACTS AND LOCATIONS:
Overall Officials: Noha A Ghallab, PhD, Study Chair — Professor of Oral Medicine & Periodontology; Ahmed I Abou- El-Fettouh, MSc, Principal Investigator — MIU; Abdelrahman Zohny, BDs, Principal Investigator — MIU; Nael M Adel, BDs, Principal Investigator — MIU; Mariam S Abdelmalak, BDs, Principal Investigator — MIU; Nesma M Shemais, PhD, Principal Investigator — Lecturer of Oral Medicine & Periodontology, Cairo University
Locations (2):
- Egypt (2):
  - International Dental Continuing Education, Cairo, Maadi
  - Faculty of Dentistry, Cairo University, Cairo, Manial

IPD SHARING:
Plan to Share IPD: No